CLINICAL TRIAL: NCT01615224
Title: Repeated Doses of Misoprostol for Treatment of Missed Abortion
Brief Title: Repeated Doses of Misoprostol for Medical Treatment of Missed Miscarriage
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: No funding
Sponsor: Kristina Gemzell Danielsson (Other)
Responsible Party: Sponsor-Investigator, Kristina Gemzell Danielsson, professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WMA11
Record Dates: First submitted 2012-06-04; First posted 2012-06-08 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-08

CONDITIONS: Missed Abortion
Keywords: missed abortion; miscarriage
MeSH Terms: conditions — Abortion, Missed; Abortion, Spontaneous | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- single dose (No Intervention): Patients receive the standard treatment with 800mcg of vaginal misoprostol
- repeated doses (Experimental): patients receive 800mcg of vaginal misoprostol. In addition to this they receive repeated doses of 400mcg oral misoprostol after 3 and 5 hours. Women of more than 9 weeks pregnancy according to last menstrual period will be given a choice of vacuum aspiration or further medical treatment with 2 additional doses of misoprostol given after 7 and 9 hours after the initial vaginal treatment.
  Interventions: Drug: misoprostol

INTERVENTIONS:
Drug: misoprostol — repeated doses of misoprostol. 400mcg of oral misoprostol given at 3, 5, 7 and 9 hours.
  Other Names: Cytotec 200mcg Pfizer
  Arms: repeated doses

SUMMARY:
Missed abortion is a condition where the fetus has perished but the miscarriage is not expelled. Women often present at a routine ultrasound or with a slight brownish discharge. Traditionally this condition has been treated with curettage or vacuum aspiration. Lately, medical treatment has become more common due to less risk of infection and other complications. The routine medical treatment is 800mcg of misoprostol administered vaginally. We wish to examine of repeated doses of 400mcg misoprostol after the initial 800mcg vaginal misoprostol increases efficacy of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age healthy no contraindication to medical treatment visible fetal structures such as yolk sac or fetus

Exclusion Criteria:

* empty gestational sac more than sparse bleeding or dilated cervix mental instability after diagnosis contraindication to medical treatment

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2012-05; Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Efficacy | 1 day
  Complete abortion as judged by ultrasound

SECONDARY OUTCOMES:
Acceptability | 1 day, 1 week, 2 weeks, 3 weeks, 5 weeks
  questionnaire on future choice of treatment method. Surgical or medical treatment if free choice. If having to have medical would she choose repeated doses or single dose?

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Gemzell Danielsson, professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Dept of Obstetrics and Gynecology, Danderyd Hospital, Stockholm, Sweden